CLINICAL TRIAL: NCT04323332
Title: A Retrospective Cohort Study to Evaluate the Efficacy and Safety of Traditional Chinese Medicine as an Adjuvant Treatment for Patients With Severe COVID-19
Brief Title: Traditional Chinese Medicine for Severe COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Hao, professor, Xiyuan Hospital of China Academy of Chinese Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020XLA015-1
Record Dates: First submitted 2020-03-08; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
Keywords: COVID-19; Traditional Chinese Medicine; Pneumonia; Coronavirus
MeSH Terms: conditions — COVID-19; Pneumonia; Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine (Experimental): TCM prescription and conventional treatments
  Interventions: Drug: Traditional Chinese Medicine Prescription
- Control (No Intervention): conventional treatments

INTERVENTIONS:
Drug: Traditional Chinese Medicine Prescription — Traditional Chinese Medicine Prescriptions have been recommended according to the Guidelines for the treatment of COVID-19 issued by National Health Commission of the PRC.
  Arms: Traditional Chinese Medicine

SUMMARY:
In December 2019, a new type of pneumonia, COVID-2019 outbroke in Wuhan ,China, and currently the infected has been reported in more than at least 75 countries.

Patients with severe COVID-19 have rapid disease progression and high mortality rate. This may attribute to the excessive immune response caused by cytokine storm. Strategies based on anti-virus drugs and treatments against symptoms have now been employed. However, these managements can't effectively treat the lethal lung injury and uncontrolled immune responses, especially in the elderly with severe COVID-19. Traditional Chinese Medicine (TCM), which treats the disease from anther perspective, has achieved satisfactory results. National Health Commission of China released a series of policies to enhance the administration of TCM prescriptions.

This study is aimed to evaluate the efficacy and safety of Traditional Chinese Medicine as an adjuvant treatment for severe COVID-19.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients were diagnosed as severe COVID-19 according to the Coronavirus disease (COVID-19) Treatment Guidance (Six edition)
2. Patients received a combined treatment of TCM and conventional therapy, or only conventional therapy.

Key Exclusion Criteria:

1. Age >85 years
2. After cardiopulmonary resuscitation
3. Patients combined with other organ failure or conditions need ICU monitoring and treatment, such as severe liver disease, severe renal dysfunction, upper gastrointestinal hemorrhage, disseminated intravascular coagulation.
4. Respiratory failure and need mechanical ventilation

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay (days) | First treatment date up to 3 months

SECONDARY OUTCOMES:
Duration (days) of supplemental oxygenation | First treatment date up to 3 months
CT imaging changes | First treatment date up to 3 months
Mortality rate | First treatment date up to 3 months
Time to Clinical Improvement (TTCI) | First treatment date up to 3 months
The pneumonia severity index scores | First treatment date up to 3 months
  The pneumonia severity index is a clinical tool helping in the risk stratification of patients with community-acquired pneumonia. It ranges from 0-395 scores and a higher score indicates higher death risk.
Time to COVID-19 nucleic acid testing negativity in throat swab | First treatment date up to 3 months
Blood immune cell count | Baseline, 7 and/ or 14 days
  Changes in leukocyte, neutral, lymphocyte counts and absolute lymphocyte count from baseline
Serum inflammatory markers | Baseline, 7 and/ or 14 days
  Changes in blood interleukin-6, c-reactive protein,SS-A/Ro antibodies and serum ferritin from baseline.
Erythrocyte sedimentation rate | Baseline, 7 and/ or 14 days
  Changes in erythrocyte sedimentation rate from baseline.
Platelet and D-dimer changes | Baseline, 7 and/ or 14 days
  Changes in platelets and D-dimers from baseline.
Creatinine changes | Baseline, 7 and/ or 14 days
  Changes in serum creatinine from baseline.
Muscle enzymes changes | Baseline, 7 and/ or 14 days
  Changes in serum muscle enzymes from baseline, including alanine aminotransferase , AST, creatine kinase, LDH.
Usage of antibiotics | First treatment date up to 3 months
  Dosing time and amounts of antibiotics；the categories of the antibiotics
Usage of glucocorticoids | First treatment date up to 3 months
  Dosing time and amounts of glucocorticoids
Frequency of adverse events | First treatment date up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hao Li, Professor, Study Chair — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Hao Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol